CLINICAL TRIAL: NCT02504749
Title: Randomised Study to Compare the Regain of Gastrointestinal Motility After General Anaesthesia Versus Spinal Anaesthesia in Caesarean Section.Kasr El Ainy,Egypt Experience
Brief Title: The Regain of Gastrointestinal Motility After General Anaesthesia Versus Spinal Anaesthesia in Caesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed El-Sharkawy, Lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KasrELAini
Record Dates: First submitted 2015-07-18; First posted 2015-07-22 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-07

CONDITIONS: G.I.T. Motility After General Versus Spinal Anaesthesia
Keywords: GIT motility; General anaesthesia; spinal anaesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: General anaesthesia group (Active Comparator): -Standard rapid sequence induction with pre-oxygenation by 100 % OXYGEN FOR 3 MINUTES FOLLOWED BY 4-5 mg/kg thiopental and 100 mg succinylcholine,cricoid pressure was applied once necessary.After correct placement of tracheal tube was confirmed,anaesthesia was maintained with up to 1.5% isoflurane and oxygen,neuromuscular blockade was maintained with 0.4 mg/kg atracurium.
  Interventions: Procedure: general anasthesia,spinal anasthesia
- Group B:Spinal anaesthesia group. (Active Comparator): Prehydration with 500 ml lactated ringer solution intravenous within 15 minutes in the sitting position.Low back was prepared and drapped in a sterile fashion with Betadine solution 10%.
  Spinal anaesthesia performed at L 2-3 or L 3-4 intervertebral space using a fine needle size 22 G.Injection of local anaesthetics into the subarachnoid space,Bupivacaine(marcaine) 1.5 -3.5 ml used.
  Interventions: Procedure: general anasthesia,spinal anasthesia

INTERVENTIONS:
Procedure: general anasthesia,spinal anasthesia — Randomization done by computer generated random number in sealed opaque envolopes.Each patient was given a study information sheet and a consent was signed. Sample size was calculated to prevent type II error. Based on these data, we would need to study 225 cases in each arm to be able to reject the null hypothesis that the rates for the experimental and control groups are equal with a probability of 80%. The type I error probability associated with this test for the null hypothesis is 0.05. We used an uncorrected chi-squared statistic to evaluate this null hypothesis. Additionally, to compensate for discontinuations, we recruited 225 women in each arm.
  450-pregnant women with an indication for caesarean section were randomly allocated .

SUMMARY:
This study aims to compare the time to regain intestinal motility after general anesthesia versus spinal anesthesia for cesarean section.

A double blinded randomized controlled trial was conducted at the Department of Obstetrics and Gynecology, Kasr El-Aini Teaching Hospital, Faculty of Medicine, Cairo University, Cairo, Egypt, between July 20 and November 20, 2015. In the study hospital, the total number of deliveries in 2012 was 15 167, 6244 (41.2%) of which were by cesarean; in 2013, the total number of deliveries was 16 057, 5200 (32.4%) of which were by cesarean.

DETAILED DESCRIPTION:
The The study protocol was approved by the Scientific Research Committee of the department. Pregnant women with indication for caesarean section were enrolled after providing informed consent. It included 450 patients who had caesarean section and were subdivided into two groups according to a randomization scale.On the day of the operation,each randomly received a closed opaque envelope for the selection of the procedure(spinal versus general).

Patients were classified into two groups:

Group A: General anaesthesia group Group B:Spinal anaesthesia group.

All patients are subjected to the following:

1. Patients admitted from the outpatient clinic at Kasr El Ainy university Maternity Hospital.
2. Explanation of the procedure to all women participating in the study.
3. Informed written consent from every woman participating in this study.
4. Full history taking:

   * Full name,age,telephone number and address.
   * Past medical history of hypertension,diabetes and other endocrine diseases,also history of abdominal operations.
   * Gravidity and parity.
5. Examination:

1-Vital signs(pulse,blood pressure,temperature and respiratory rate). 2-Measurement of weight in kilograms,height in meters and calculation of body mass index.

6-Full laboratory investigations especially Complete blood count,liver functions,kidney functions,coagulation profile and random blood sugar.

7-Ultrasound assessment of fetal well being.

8-All women fasting for at least 8 hours prior to surgery.

General anaesthesia steps:

-Standard rapid sequence induction with pre-oxygenation by 100 % OXYGEN FOR 3 MINUTES FOLLOWED BY 4-5 mg/kg thiopental and 100 mg succinylcholine,cricoid pressure was applied once necessary.After correct placement of tracheal tube was confirmed,anaesthesia was maintained with up to 1.5% isoflurane and oxygen,neuromuscular blockade was maintained with 0.4 mg/kg atracurium.

Spinal anaesthesia steps:

Prehydration with 500 ml lactated ringer solution intravenous within 15 minutes in the sitting position.Low back was prepared and drapped in a sterile fashion with Betadine solution 10%.

Spinal anaesthesia performed at L 2-3 or L 3-4 intervertebral space using a fine needle size 22 G.Injection of local anaesthetics into the subarachnoid space,Bupivacaine(marcaine) 1.5 -3.5 ml used.

Operative data:

* Caesarean section done by senior resident.
* Skin opened by pfannensteil incision
* The abdomen opened in layers.
* The peritoneum opened by elevating it with two clamps placed 2 cm apart. It is incised sharply superiorly to the upper pole of the incision and downward to just above bladder reflection.
* The lower peritoneal flap elevated and gentle blunt bladder dissection done.
* Transverse incision of the lower uterine segment.
* The baby is delivered:a hand is slipped into the uterine cavity between the symphysis and fetal head.Head elevation with the fingers and palm through the incision.
* Intravenous infusion containing 20 units of oxytocin after shoulder delivery.
* Spontaneous placental delivery.
* Closure of uterine incision in two layers using blunt needle and absorbable continuous Vicryl 1 sutures (Ethicon; Somerville,New Jersey,, USA) in a continuous double layer.
* Closure of visceral and parietal peritoneum by continuous absorbable suture Vicryl 2-0.
* Rectus sheath sutured using continuous absorbable suture Vicryl 1 sutures.
* In all patients, the fascia was closed with continuous Vicryl 1 sutures, subcutaneous fat was closed with interrupted Vicryl 2-0 sutures, and the skin was closed with subcuticular Prolene 2-0 sutures (Ethicon).

The data were recorded including presence of adhesions,application of intraperitoneal towels,estimated blood loss,operative time,time from start of caesarean section to fetal extraction and closure events.

After the end of surgery:

* close observation for vital data,vaginal bleeding and urine output.
* The same hospital fluid regimen with 500 ml of 5 % glucose every 6 hours,500 ml of ringer every 12 hours and 500 ml saline every 24 hours.
* Postoperatively, all patients were given 75 mg diclofenac sodium (Voltaren; Novartis,Cairo, Egypt) as intravenous infusion in dextrose, followed by 50 mg diclofenac potassium (Cataflam; Novartis) orally every 8 hours for pain relief.
* No oral or rectal bowel stimulants were given after surgery.
* Auscultation of intestinal sounds started two hours after operation and was performed at one hour interval till normal bowel sounds were detected.
* The patients allowed to sip small amount of water only 12 hours postoperatively.
* The oral intake of clear fluid and soft food was allowed when normal bowel sounds were detected and flatus has passed with advancement to regular diet after passage of first bowel motion.
* Clinically significant ileus was considered with appearance of group of manifestations(persisting more than 24 hours or requiring nasogastric tube placement) which include absent or hypo active bowel sounds,abdominal distension and more than three episodes of vomiting with or without crampy abdominal pain.
* Eligible criteria for hospital discharge included:stable vital signs with no febrile morbidity for at least 24 hours,ability to ambulate and to urinate without assistance,passage of bowel motion,ability to tolerate solid food without emesis and absence of unresolved other postoperative complications.

The main outcome measures are:

* Case number
* Age
* Parity
* Gestational age
* Body mass index.
* Duration of surgery.
* Time of 1 st intestinal sound
* Time of 1 st flatus.
* Time of 1 st motion
* Duration of hospital stay.
* Post operative fever,distension or ileus.
* Opioid and Non steroidal anti-inflammatory use.

ELIGIBILITY:
Inclusion Criteria:

* Patients set for planned cesarean section under general or spinal anesthesia:

  1. age from 18 to 37 years.
  2. Full term(37-41 weeks).
  3. Singleton pregnancy.
  4. Hemoglobin level more than 11 gm/dl.

Exclusion Criteria:

1. Contraindication to regional anesthesia i.e(patient refusal,coagulopathy,significant hypovolemia,systemic or local sepsis,increased intracranial pressure,severe stenotic valvular heart disease,pre existing neurologic conditions and local anesthetic or fentanyl allergy.
2. High risk pregnancies as pre eclampsia,eclampsia,any medical disorder(DM,cardiac and thyroid diseases).
3. Previous intestinal surgery,previous C.S. and previous gynecological operations.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Time of first flatus | 3 months

SECONDARY OUTCOMES:
postoperative complications | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kasr El Ainy, Study Chair — Office Dean
Locations (1):
- Mohamed Abdel Aziz El Sharkawy, Cairo, Egypt